CLINICAL TRIAL: NCT06612632
Title: A Umbrella Study to Evaluate the Safety and Preliminary Efficacy of Combined or Sequential Immunotherapy in Patients with Advanced Solid Tumors Progressing on Clinical Trial Drugs
Brief Title: Immunotherapy Rechallenge in Patients with Solid Tumors in Clinical Trials
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, NING_LI, professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC20231105
Record Dates: First submitted 2024-07-14; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-07

CONDITIONS: Cancer
Keywords: immunotherapy; rechallenge; clinical trail; solid tumor
MeSH Terms: conditions — Neoplasms | interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: An Umbrella Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Combination therapy (Experimental): Research drug in combination with Toripalimab
  Interventions: Drug: research drug in combination with Toripalimab
- Sequential therapy (Experimental): Toripalimab
  Interventions: Drug: Toripalimab
- RWS cohort (No Intervention): observation

INTERVENTIONS:
Drug: research drug in combination with Toripalimab — research drug in combination with Toripalimab
  Arms: Combination therapy
Drug: Toripalimab — Toripalimab
  Arms: Sequential therapy

SUMMARY:
This study plans to include approximately 60-100 patients with advanced solid tumors who have progressed on clinical trial drugs. It will use an open-label, single-arm, multi-cohort umbrella design. In the first phase, patients who have progressed during treatment with novel tumor immunotherapy drugs will initially be targeted, combining or sequencing with PD-1 monoclonal antibody therapy. The inclusion criteria for frontline clinical trials are as follows: priority will be given to phase I clinical trials of novel immunotherapeutics as monotherapy, such as tumor vaccines, NK cell therapy, and new immune checkpoint inhibitors. Based on preliminary data, these have shown synergistic effects with PD-1/L1 monoclonal antibodies. In principle, the same investigational drug will only be used in either a combination or sequencing cohort. Subsequently, the study will expand to include patients who have progressed on other clinical trial treatments, combining or sequencing with other immune mechanism drugs.

DETAILED DESCRIPTION:
This study plans to include approximately 60-100 patients with advanced solid tumors who have progressed on clinical trial drugs, using an open-label, single-arm, multi-cohort umbrella design. In the first phase, patients who have progressed during treatment with novel tumor immunotherapy drugs will initially be targeted, combining or sequencing with PD-1 monoclonal antibody therapy. The selection criteria for frontline clinical trials are as follows: priority will be given to phase I clinical trials of novel immunotherapeutics as monotherapy, such as tumor vaccines, NK cell therapy, and new immune checkpoint inhibitors. Based on preliminary data, these have shown synergistic effects with PD-1/L1 monoclonal antibodies. In principle, the same investigational drug will only be used in either a combination or sequencing cohort. Subsequently, the study will expand to include patients who have progressed on other clinical trial treatments, combining or sequencing with other immune mechanism drugs.

Based on the interventions, the study is divided into combination therapy cohorts, sequential therapy cohorts, and real-world cohorts. The combination therapy cohorts will be further subdivided according to the investigational drug the patients received in the frontline setting: for instance, patients who have progressed on investigational drug A (e.g., SG1827) will receive drug A combined with PD-1 monoclonal antibody therapy (cohort A), and patients who have progressed on investigational drug B (e.g., ABO2011) will receive drug B combined with PD-1 monoclonal antibody therapy (cohort B), and so on. In the sequential therapy cohorts, regardless of the investigational drug used in the frontline setting, patients will receive PD-1 monoclonal antibody therapy. The real-world cohorts will include patients who do not meet the inclusion criteria for the aforementioned cohorts or refuse to participate in the interventional trials, with only subsequent treatment information, tumor progression, and overall survival being collected.

No specific sample size is predetermined for each cohort, and the study team may adjust the cohort sizes based on preliminary study results. In the combination therapy cohorts, the dosage and administration method of the investigational drugs will continue as per the patients' previous trial treatments. In both the combination and sequential therapy cohorts, the PD-1 monoclonal antibody will be administered at a fixed dose of 200 mg every 21 days or 3 mg/kg every 14 days. The treatments will continue until disease progression, death, or the occurrence of intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent or metastatic solid tumors confirmed by histopathology that cannot be treated with curative local therapy
2. Prior systemic anti-tumor treatment requirements: Previous first-line treatment involved a clinical trial of a new drug, with disease progression, and deemed by the investigator to no longer benefit from it
3. Suggested first dose administered within 12 weeks after the last treatment.
4. According to the RECIST 1.1 criteria, there should be at least one measurable lesion or more
5. ECOG PS 0-2 points
6. expected survival ≥ 3 months
7. as assessed by the investigator, major organ functions are good enough and can tolerate the experimental treatment regimen used in this study
8. subjects can understand and comply with the study procedures, sign the informed consent form, and voluntarily participate in this study
9. patients included in the real-world cohort who do not meet the aforementioned inclusion criteria or refuse to participate in the aforementioned interventional experimental treatment

Exclusion Criteria:

1. Previous exposure to immunotherapy (standard treatment or clinical trials) resulted in severe immune-related adverse events, as assessed by the investigator, making the re-administration of immunotherapy inappropriate.
2. Previous adverse reactions to advanced solid tumors have persisted, and the investigator anticipates these might impact the safety evaluation of the investigational drug
3. Previously experienced hyperprogression during immune therapy (conventional treatment or clinical trials), and the Other conditions deemed unsuitable for participation in this study by the investigator believes that no further benefit can be gained from this study. Criteria include: (1) Tumor progression time less than two months during immunotherapy
4. (2) Tumor burden increased by over 50% compared to baseline
5. (3) Tumor growth rate post-immunotherapy exceeds twice the previous rate
6. Central nervous system metastases or leptomeningeal metastases with clinical symptoms
7. During the screening period, subjects are determined by the investigator to have severe or uncontrolled underlying diseases (such as hypertension, diabetes, cardiovascular diseases, pulmonary diseases, autoimmune diseases, etc.)
8. Received other anti-tumor therapy between the last front-line therapy and the first dose of the study drug
9. Other conditions deemed unsuitable for participation in this study by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing AEs | 5 years
  Number of participants with AE by CTCAE v5.0.
Number of Participants Experiencing TEAEs | 5 years
  Number of Participants with TEAEs by CTCAE v5.0.
Number of Participants Experiencing TRAEs | 5 years
  Number of Participants with TRAEs by CTCAE v5.0.
Number of Participants Experiencing SAEs | 5 years
  Number of Participants with SAEs by CTCAE v5.0.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 5 years
  Overall Response Rate (ORR)
Disease Control Rate(DCR) Disease Control Rate(DCR) Disease Control Rate(DCR) Disease Control Rate(DCR) | 5 years
  Disease Control Rate(DCR)
Duration of Response (DOR) | 5 years
  Duration of Response (DOR)
Progression-Free Survival (PFS) | 5 years
  Progression-Free Survival (PFS)
Overall Survival (OS) | 5 years
  Overall Survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Academic papers publishing research results